CLINICAL TRIAL: NCT03804723
Title: Glucocorticoids Withdrawal in Early Systemic Lupus Erythematosus: a Randomized Placebo-controlled Equivalence Trial
Brief Title: Glucocorticoids Withdrawal in Early Systemic Lupus Erythematosus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Marta Mosca, Assistant Professor of Rheumatology, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Systemic Lupus Erythematosus; Glucocorticoids; Therapy Withdrawal
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: This is a 36 month, randomized, double-blind, placebo-controlled, parallel-groups, equivalence multicenter trial in patients with inactive SLE to evaluate if low disease activity can be sustained with withdrawal of glucocorticoids
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GC withdrawal (Experimental)
  Interventions: Drug: oral Prednisone 5mg
- non GC withdrawal (Placebo Comparator)
  Interventions: Drug: oral Prednisone 5mg

INTERVENTIONS:
Drug: oral Prednisone 5mg — patients randomized to this arm will stop prednisone 5 mg

SUMMARY:
This is a 36 months, randomized, double-blind, placebo-controlled, parallel-groups, equivalence multicenter trial in patients with inactive Systemic Lupus Erythematosus to evaluate if low disease activity can be sustained with withdrawal of glucocorticoids in patients on stable clinical remission or low disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE according to the EULAR/ACR criteria within three years from screening visit
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information in accordance with national subject privacy regulations
* Aged 18 to 75 years old, inclusive, at the time of informed consent
* Documented diagnosis of SLE according to the current ACR criteria
* Stable immunosuppressive treatment for SLE for a minimum of one year/six months
* Stable treatment with antimalarials for a minimum of 3 months
* stable (lasting for at least 6 months) low disease activity

Exclusion Criteria:

* Disease activity (non LLDAS) within 6 months prior to screening
* Concomitant ongoing conditions (e.g. asthma, Crohn's disease) that require treatment with systemic GC (excluding topical or inhaled GC).
* Unwillingness or inability to comply with the requirements of this protocol, including the presence of any condition (physical, mental, social) likely to affect the subject returning for follow-up visits on schedule
* Nursing mothers, pregnant women or women planning to become pregnant during the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
disease flare | 35 months
  The primary endpoint is the proportion of patients who will experience a disease during the follow-up period in the groups given prednisone 5 mg or placebo in the double-blind period.

IPD SHARING:
Plan to Share IPD: Undecided